CLINICAL TRIAL: NCT05319990
Title: Pathogenesis of Kidney Disease in Type 1 Diabetes: a Modern Kidney Biopsy Cohort (The PANDA Study)
Acronym: PANDA
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 22-0250
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes; Diabetic Kidney Disease; Diabetes Complications; Diabetic Nephropathies; Autoimmune Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies; Diabetes Complications | interventions — p-Aminohippuric Acid; Iohexol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the study, the investigators will collect blood, urine, and tissue samples for assessment of kidney function and kidney injury markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PANDA, T1D: New participants with T1D will be enrolled at the University of Colorado and University of Washington.
- PANDA Sub Study, Former CROCODILE Participants: Participants will be enrolled from the existing CROCODILE study (COMIRB # 19-1282), adding longitudinal follow-up to completed kidney biopsies and baseline data and biosample acquisition.
  Interventions: Drug: Aminohippurate Sodium Inj 20% Diagnostic aid/agent used to measure effective renal plasma flow (ERPF); Drug: Iohexol Inj 300 MG/ML Diagnostic aid/agent used to measure glomerular filtration rate (GFR)

INTERVENTIONS:
Drug: Aminohippurate Sodium Inj 20% Diagnostic aid/agent used to measure effective renal plasma flow (ERPF) — PAH (Basic Pharma, Geleen, Netherlands) has been used to measure ERPF in human research for 7 decades, and is very well tolerated and generally recognized as safe with low toxicity.
  Other Names: Sodium 4-amino hippurate (PAH) inj 20% 2g/10mL; Para-aminohippurate
  Groups: PANDA Sub Study, Former CROCODILE Participants
Drug: Iohexol Inj 300 MG/ML Diagnostic aid/agent used to measure glomerular filtration rate (GFR) — Iohexol (Omnipaque 300, GE Healthcare, Chicago, IL) is a nonionic, low osmolar contrast agent with a history of extensive use in Radiology practice (for contrast x-rays) that shares many qualities of an ideal GFR marker, like inulin, such as not being absorbed, metabolized, or secreted by the kidney.
  Other Names: omnipaque 300
  Groups: PANDA Sub Study, Former CROCODILE Participants

SUMMARY:
Diabetic kidney disease (DKD) occurs in up to 40% of people with type 1 diabetes (T1D), often leading to kidney failure and markedly magnifying risks of cardiovascular disease and premature death. Landmark T1D kidney biopsy studies identified the classic pathological lesions of DKD, which have been attributed largely to hyperglycemia. Recent advances in continuous glucose monitoring (CGM) and automated insulin delivery have facilitated improved glycemic control, but the residual risk of DKD continues to be high. In addition, obesity and insulin resistance (IR) have accompanied intensive glycemic therapy and may promote mitochondrial dysfunction and inflammation. Deciphering the molecular underpinnings of DKD in modern-day T1D and identifying modifiable risk factors could lead to more effective and targeted therapies to prevent DKD.

DETAILED DESCRIPTION:
The overall goal of this project is to characterize the molecular, morphometric, and metabolic features of DKD over the modern clinical course of T1D. The investigators hypothesize that perturbed kidney energetics and hypoxia are central metabolic pathways in the development of DKD. Kidney hypoxia stems from a mismatch between increased renal energy demand (e.g., increased glomerular filtration rate [GFR] and tubular reabsorption of sodium) and impaired substrate metabolism (e.g., IR and mitochondrial dysfunction) and results in activation of the hypoxia-inducible factor (HIF) system. Although upregulation of HIF1α confers favorable short-term effects, sustained activation promotes cellular injury. Supporting these hypotheses, data from our group and others have shown that obesity, IR, and The investigators also found that youth with T1D exhibit kidney hypoxia by MRI that strongly associates with IR and mitochondrial dysfunction. Moreover, our preliminary single-cell RNA sequencing (scRNA-seq) data from kidney biopsies demonstrate upregulated tubular expression of HIF1α in adults with T1D vs. healthy controls. The investigators propose to build a unique new longitudinal kidney biopsy cohort (N=100) spanning the critical duration of T1D over which DKD initiates and progresses (5-30 years). Participants will be enrolled from our existing CROCODILE study (adding longitudinal follow-up to completed kidney biopsies and baseline data and biosample acquisition) and from new enrollment at the University of Colorado and University of Washington. Normative kidney biopsy data will be provided from our existing cohort of healthy controls (N=20) and the Kidney Precision Medicine Project (KPMP). The investigators will implement state-of-the-art molecular (scRNA-seq) and morphometric interrogation of kidney tissue and rigorous metabolic phenotyping to include kidney magnetic resonance imaging (MRI), direct measurements of glycemia (continuous glucose monitoring), intraabdominal fat (dual-energy X-ray absorptiometry), estimation of insulin sensitivity by a T1D-validated equation, and (in a subset) GFR (iohexol clearance) and renal plasma flow (p-aminohippurate clearance). Participants will be followed longitudinally for DKD outcomes. A subset of 20 participants will undergo repeat kidney biopsies and associated procedures 3 years after baseline kidney biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at enrollment (rationale: this study focuses on determinants of early DKD over the course of T1D in adults)
* T1D duration >5 years (rationale: DKD in T1D rarely manifests prior to 5 years of disease duration)
* HbA1c <11% (rationale: HbA1c ≥ 11% exceeds the average HbA1c at most academic center and would limiting the generalizability of our study findings)

Exclusion Criteria:

* T2D and monogenic diabetes (rationale: our study focuses on T1D)
* Recent diabetic ketoacidosis, i.e., <1 month (rationale: safety and insulin resistance and tubular dysfunction of DKA can confound study findings)
* eGFR < 30 ml/min/1.73m2 or dialysis treatment (rationale: to reduce the likelihood of identifying secondary pathways that are not specific to kidney injury from T1D)
* Kidney transplant recipients (rationale: molecular confounding from immunosuppression)
* Kidney biopsy contraindications (rationale: safety - kidney biopsy):

  * Evidence of bleeding disorder or complications from bleeding
  * Use of aspirin, Nonsteroidal anti-inflammatory drugs (NSAIDS) or other blood thinner that cannot be safely stopped for a sufficient time before and after the biopsy to avoid additional risk of bleeding.
  * INR > 1.4
  * Hemoglobin (Hgb) < 10 mg/dL (Colorado) [altitude]
  * Hemoglobin (Hgb) < 9 mg/dL (Washington)
  * Platelet count < 100,000 / µL
  * Uncontrolled or difficult to control hypertension (> 150/90 mmHg at the day of biopsy)
  * Single kidney (either by history, documented by prior imaging or ultrasound performed prior to the biopsy)
  * Kidney size: One or both kidneys < 8 cm
  * Hydronephrosis or other important renal ultrasound findings such as significant stone disease
  * Any evidence of a current urinary tract infection as indicated on day of biopsy
  * Clinical evidence of non-diabetic renal disease
  * Positive urine pregnancy test or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators propose to address the specific aims of this study in a cross-sectional project with 70 newly enrolled adults with T1D and 30 former CROCODILE participants (COMIRB #19-1282).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Renal Oxygenation | 30 min
  Blood oxygen level dependent (BOLD) MRI
Renal Perfusion | 30 min
  Arterial Spin Labeling (ASL) MRI
Insulin Sensitivity | 4.5 hours
  Hyperinsulinemic-Euglycemic Clamp

SECONDARY OUTCOMES:
Glomerular Filtration Rate (GFR) | 3 hours
  Iohexol Clearance Study
Effective Renal Plasma Flow (ERPF) | 2.5 hours
  PAH Clearance Study

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided